CLINICAL TRIAL: NCT00310674
Title: A Phase III, Single Center, Open Label, Uncontrolled Study to Evaluate the Immunogenicity, Safety and Tolerability, of the Chiron Meningococcal C Conjugate Vaccine When Administered to Healthy Premature and Non Premature Children at 3, 5, 11 Months of Age Concomitantly With a Hexavalent Infant Vaccine
Brief Title: Immunogenicity, Safety and Tolerability, of Chiron Meningococcal C Conjugate Vaccine Administered to Healthy Premature and Non Premature Children of 3 Months of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Novartis Vaccines (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: M14P3; Impact N° 926
Record Dates: First submitted 2006-04-03; First posted 2006-04-04 (Estimated); Last update posted 2007-03-13 (Estimated); Status verified 2007-03

CONDITIONS: Prevention of Meningococcal Infection
Keywords: Prevention of Meningococcal Meningitis; meningococcal vaccines; conjugate; Immunology; infant
MeSH Terms: interventions — serogroup C meningococcal conjugate vaccine

INTERVENTIONS:
Biological: Meningococcal C Conjugate Vaccine

SUMMARY:
Immunogenicity, Safety and Tolerability, of Chiron Meningococcal C Conjugate Vaccine Administered to Healthy Premature and Non Premature Children of 3 months of age

ELIGIBILITY:
Inclusion Criteria:

* Healthy children of 11 to 15 weeks of age

Exclusion Criteria:

* Children who previously received any kind of Meningococcal C vaccine, DTaP-IPV-HBV-Hib vaccine or a Hepatitis B vaccine at birth
* Children who have a previous ascertained or suspected disease caused by N. meningitidis, Corynebacterium diphtheriae, Clostridium tetani, poliovirus, Hepatitis B or H. influenzae type b, culture proven Bordetella pertussis, or clinical condition of spasmodic cough for a period longer than or equal to 2 weeks associated with apnea or whooping
* Children who have had household contact with and/or intimate exposure to an individual with culture proven N. meningitidis serogroup C or Bordetella pertussis, within the previous 60 days

Ages: 11 Weeks to 15 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150
Dates: Start 2004-09

PRIMARY OUTCOMES:
antibody response, as measured by ELISA, to N. meningitidis serogroup C at one month following three doses of MenC Conjugate Vaccine administered at 3, 5, 11 months of age, together with a hexavalent vaccine.
safety and tolerability

SECONDARY OUTCOMES:
antibody response as measured by ELISA at 1 month after second dose of MenC Vaccine and before third dose with hexavalent vaccine
antibody response as measured by BCA in subset of subjects in each group, at 1 month after second dose, immediately before the third and at 1 month following the third dose of MenC Vaccine together with a hexavalent vaccine.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis - Information Services, Principal Investigator — Novartis Vaccines & Diagnostics
Locations (1):
- Istituto di Pediatria, Università degli Studi di Milano, Milan, Italy